CLINICAL TRIAL: NCT05308914
Title: Self-Management and Resilience Trajectories in African American Adults With Hypertension
Status: Completed | Type: Observational
Sponsor: Case Western Reserve University (Other)
Collaborators: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Carolyn Still, Assistant Professor, Case Western Reserve University
Other Study IDs: 1R21NR020489-01A1 (NIH)
Record Dates: First submitted 2022-03-09; First posted 2022-04-04 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Hypertension; Self-Management; Quality of Life; Compliance, Medication; Compliance, Treatment; Compliance, Patient
Keywords: Hypertension; Self-Management; Resilience
MeSH Terms: conditions — Hypertension; Medication Adherence; Patient Compliance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: None Retained — Specimens: Blood will be obtained at baseline, 3 months, and 6 months. Subjects will have blood samples (2 tubes, 1 teaspoon=5 ml each tube) drawn for Interleukin 6 (IIL-6) and High sensitivity C-reactive Protein (CRP) and cortisol serum to assess (~10 minutes to complete).
  Hair samples will be obtain at baseline and 6 months for Cortisol Concentration
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Resilience Study Cohort: Observational, descriptive longitudinal cohort design. See inclusion and exclusion criteria for more information

SUMMARY:
Hypertension (HTN) rates have increased worldwide, but the most significant increase in the incidence of morbidity and mortality has been in African Americans (AA)1,2 (43% vs 27% for other U.S. population groups). Despite evidence of positive benefits from lifestyle modification (healthy diet, reduced sodium intake, increased physical activity, smoking cessation) and prescribed antihypertensive therapy (AHT) many AA with HTN do not adhere to their treatment regimens. Consistent, effective lifelong self-management is required to sustain optimal BP control and thus reduce morbidity and mortality. Self-managing HTN to a blood pressure (BP) <130/80 mm Hg presents challenges such as juggling multiple medications and health care providers, dealing with complex recommendations and treatment regimens, and coping with negative emotional states. Few studies have examined the biopsychosocial mechanisms that foster effective HTN self-management and resilience among AA living with HTN. Understanding the mechanisms that influence HTN self-management and resilience in AA holds the promise of new modifiable targets for behavior-change interventions.

This study explores the relationship among resilience precursors on hypertension (HTN) self-management behaviors, stress response, and the effects that these relationships have on health outcomes-health-related quality of life (HRQOL) and blood pressure (BP) in African Americans (AA) with HTN over a 6-month period.

DETAILED DESCRIPTION:
This study identifies profiles of self-management and the resilience trajectories in AA with HTN can lead to culturally appropriate, patient-centered interventions that improve their HTN self-management, quality of life, and long-term compliance.

This study aims to:

1. Assess the association among resilience precursors (dispositional optimism and resilience, emotion regulation); stress response (physiological: cortisol, interleukins [IL-6] and psychological: depression cognitions, perceived stress); hypertension self management behaviors (self-efficacy for chronic disease management, medication adherence to antihypertensives); and health outcomes (HQROL and BP) in AA with HTN at baseline and months 3 and 6.
2. Determine if stress response mediates the relationship between resilience precursors and health outcomes over time when controlling for risk regulators.
3. Determine if self-management behaviors mediates the relationship between resilience precursors and health outcomes over time when controlling for risk regulators.
4. Identify resilience trajectory patterns and factors that influence HTN self-management behaviors over time.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as African American
* 25 years of age or older
* Diagnosed with hypertension and prescribed one antihypertensive medication
* BP >130/80 mmHg
* Have at least one additional chronic health conditions
* Able to read/understand English

Exclusion Criteria:

* Unable to give informed consent or judged to have impaired cognitive ability or severe memory
* Have experienced a major CVD event or procedure (e.g., myocardial infarction, stroke, heart surgery) within the past year

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants self-identify as African American, 25 years and older, who have a diagnosis of hypertension and living in the Greater Cleveland area.
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
systolic and diastolic Blood Pressure | Baseline - 6 months
  Measure of participants' in clinic blood pressure (average of three blood pressure readings).
PROMIS Global Health-10 [health-related quality of life] | Baseline - 6 months
  Total summed score on PROMIS Global Health-10 that range from 4-20.Higher scores indicate greater health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Still, PhD, Principal Investigator — Case Western Reserve University, School of Nursing
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided